CLINICAL TRIAL: NCT00798460
Title: A Multicenter, Randomized, Controlled Tial of Combination Therapy for Lamivudine-resistant Chronic Hepatitis B Patient: Comparing Clevudine Plus Adefovir With Lamivudine Plus Adefovir
Brief Title: Efficacy of Clevudine Plus Lamivudine for Lamivudine-resistant Chronic Hepatitis B Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: could not enroll patients
Sponsor: Inje University (Other)
Collaborators: Bukwang Pharmaceutical (Industry)
Responsible Party: June Sung Lee, Ilsanpaik hospital, Inje University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB-0809-055
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic hepatitis B; lamivudine resistance; clevudine
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — adefovir; adefovir dipivoxil; clevudine; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lamivudine plus adefovir (Active Comparator)
  Interventions: Drug: adefovir; Drug: lamivudine
- Clevudine plus adefovir (Active Comparator)
  Interventions: Drug: adefovir; Drug: clevudine

INTERVENTIONS:
Drug: adefovir — adefovir 10mg
  Other Names: Hepsera
Drug: clevudine — clevudine 30mg
  Other Names: Levovir
  Arms: Clevudine plus adefovir
Drug: lamivudine — lamivudine 100mg
  Other Names: Zeffix
  Arms: Lamivudine plus adefovir

SUMMARY:
The purpose of this study is to determine the optimal antiviral treatment for lamivudine resistant hepatitis B patients.

DETAILED DESCRIPTION:
Lamivudine with adefovir combination therapy has been known as effective antiviral therapy for lamivudine resistant chronic hepatitis B patients. It is superior to adefovir monotherapy since the incidence of viral breakthrough of combination therapy used to be less than that of adefovir monotherapy in lamivudine resistant chronic hepatitis B patients. Clevudine, which is being marketed in Korea, is a nucleoside analogue of the unnatural beta-L configuration that has potent activity against HBV. It has demonstrated potent antiviral efficacy and significant biochemical improvement after 24 weeks of therapy. We hypothesized that clevudine plus adefovir combination therapy for lamivudine resistant patients might be as effective as the lamivudine plus adefovir combination therapy.

In detail, we designed to perform this clinical study comparing the combination of clevudine and adefovir with lamivudine plus adefovir in lamivudine resistant chronic hepatitis B patient. Total treatment duration of both groups will be 12 months, and compare the efficacy of antiviral effects of these drugs.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg positive and anti-HBs negative more than 6 months
* YMDD mutation (+)during lamivudine therapy
* Serum ALT more than two times upper normal value

Exclusion Criteria:

* HAV IgM Ab + and/or HCV Ab+ and/or HDV Ab and/or HIV Av+
* The sign of decompensated liver disease
* Pregnant or lactating woman
* The history of hemoglobinopathy, autoimmune hepatitis, alcoholic liver disease
* Hemoglobin less than 8 g/dL (male), 7.5g/dL (female) or neutrophil count less than 1500/mm3 or platelet count less than 50,000/mm3
* Serum creatinine more than 1.5 times upper normal limit value
* The sign of malignancy or suggestive of malignancy or the history of malignancy, the recurrence rate within 2 years of which is more than 20%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-12; Primary Completion 2010-06 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
HBV DNA titer < 300 copies/mL | 48 week

SECONDARY OUTCOMES:
Normalization of serum ALT, loss of HBeAg and HBsAg, incidence of adefovir resistance | 48 week

CONTACTS AND LOCATIONS:
Overall Officials: June Sung Lee, M.D., Principal Investigator — Department of Internal Medicine, Ilsanpaik hospital, Inje Univeristy, 2240 Daewha-dong, Ilsanseo-gu, Goyang, Gyunggi, Korea, 411-706
Locations (1):
- Ilsanpaik hospital, Goyang, Gyunggi, South Korea